CLINICAL TRIAL: NCT02862899
Title: Use of a Heating Cable to Obtain Hyperthermia During Intraperitoneal Chemotherapy
Acronym: CHIPOFIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORTEGA 2012
Record Dates: First submitted 2016-08-05; First posted 2016-08-11 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intraperitoneal Chemotherapy

ARMS (1):
- Heating cable (Experimental)
  Interventions: Device: Thermowire

INTERVENTIONS:
Device: Thermowire
  Other Names: Heating cable

SUMMARY:
The investigator will study the possibility of in situ heating of the liquid containing the chemotherapy, so as to avoid the need for an external pumping system with its complexity, and its associated risks and costs.

The use of a heating cable (prototype hereinafter called Thermowire, made by the company EFS, which is in charge of its development) was patented and tested in pigs in two studies that included 15 animals altogether (in 7 of which the heating cable was used). The aim of the first study was the purely safety aspects, while the efficacy to obtain hyperthermia, the quality and the homogeneity of the hyperthermia and its effect on the tissue penetration of the chemotherapy were evaluated in a second study. The results obtained justify transfer to use in humans in the context of a clinical trial so as to obtain CE certification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with national health insurance cover
* With scheduled hyperthermic intraperitoneal chemotherapy (HIPEC) because of known peritoneal disease (primary or secondary)
* Who have provided written consent

Exclusion Criteria:

* Persons under guardianship
* Persons under 18 years old
* Pregnant or breast-feeding women
* Allergy to latex
* Abandon of HIPEC following surgical exploration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
SAE due to use of Thermowire | Through study completion up to 22 months
  In particular visceral thermal lesions or electric accidents.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Ortega-Deballon P, Facy O, Binquet C, Delroeux D, Rat P. CHIPOFIL: A pilot study assessing the feasibility of HIPEC without extracorporeal circuit. Pleura Peritoneum. 2019 Jul 26;4(3):20190008. doi: 10.1515/pp-2019-0008. eCollection 2019 Sep 1. PMID 31667330